CLINICAL TRIAL: NCT07306975
Title: Comparative Analysis of SUV Measurements Using Different Correction Methods in Oncological PET/CT Imaging.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Kamel Hamed Ahmed, Resident doctor, Assiut University
Other Study IDs: SUV measurements in PET/CT
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cancer Patients Referred to do PET/CT Study
Keywords: SUV measurements , correction, PET/CT
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: PET/CT with 18-FDG — * Patients will fast for at least 4 hrs before imaging with blood glucose level (<200 mg/dl) before intravenous administration of F18-FDG.
  * Imaging will be performed approximately 45 to 60 min after 18F-FDG injection, an imaging field of view from the base of skull to mid-thighs with the arms above the head whenever possible is used or otherwise the arms are positioned beside the body.

SUMMARY:
-To measure SUVs by using different correction methods in oncological PET/CT imaging.

DETAILED DESCRIPTION:
-To compare between SUV measurements in the tumor and liver using different standardizing parameters such as: body weight, lean body mass and body surface area.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients (> 18 years old) referred to nuclear medicine unit to do F18-FDG PET/CT study.

Exclusion Criteria:

* Patients < 18 years old.
* Patients with increased FDG uptake on tissue associated with non-malignant causes such as diffuse bone marrow FDG uptake or inflammatory.
* Patients with extensive metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Cancer patients (> 18 years old) referred to nuclear medicine unit to do F18-FDG PET/CT study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
-To measure SUVs by using different correction methods in oncological PET/CT imaging. | 1/12/2025 to 1/10/2027
  -To compare between SUV measurements in the tumor and liver using different standardizing parameters such as: body weight, lean body mass and body surface area.

SECONDARY OUTCOMES:
To determine if SUVbsa is more accurate than SUVbw in obese patients. | 1/12/2025 to 1/10/2027
  -To determine if ''normalization of FDG uptake for the body surface area'' (SUVbsa) is independent of the patient's body size and is more reliable than SUVbw.

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Gamal Eldin Mostafa, Professor, doctor, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Result] Kim CK, Gupta NC, Chandramouli B, Alavi A. Standardized uptake values of FDG: body surface area correction is preferable to body weight correction. J Nucl Med. 1994 Jan;35(1):164-7. PMID 8271040
- [Result] Nakaichi T, Funamoto K, Yamashita S, Yamamoto H, Yokoyama K. Clinical Usefulness of Standardized Uptake Value Normalized to Lean Body Mass Measured Using a Body Composition Analyzer. Cureus. 2025 May 30;17(5):e85089. doi: 10.7759/cureus.85089. eCollection 2025 May. PMID 40589668
- [Result] Azmi NHM, Suppiah S, Liong CW, Noor NM, Said SM, Hanafi MH, et al. Reliability of standarized uptake value normalized to lean body mass using the liver as a reference organ, in contrast-enhanced 18F-FDG PET/CT imaging. Radiography. 2018;24(2):112-117. doi:10.1016/j.radi.2017.09.006.
- [Result] Ahmed A, Ali M, Salah H, Eisa RE, Mohieldin H, Omer H, et al. Evaluation of uptake values of FDG: Body surface area Vs. body weight correction. Radiat Phys Chem. 2022;201:110482. doi:10.1016/j.radphyschem.2022.110482 .